CLINICAL TRIAL: NCT06793540
Title: Effectiveness of Self-posturotherapy on the Elimination of Residual Fragments After Treatment of Lower Calyx Urinary Stones by Extracorporeal Lithotripsy or Retrograde Flexible Ureteroscopy.
Acronym: ALUR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-06-024-ALMERAS(ALUR); 2024-A02267-40 (Other: Numéro ID RCB ( ANSM))
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Stone, Kidney
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Model Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self-posturotherapy (Experimental): standard care (according to recommendations) + self-posturotherapy program
  Interventions: Behavioral: SELF POSTUROTHERAPIE
- Standard care (No Intervention): standard care alone (according to recommendations)

INTERVENTIONS:
Behavioral: SELF POSTUROTHERAPIE — a simplified posturotherapy protocol that can be carried out by the patient himself. This protocol is based on the same principles as posturotherapy carried out by a physiotherapist by combining inclined positioning, percussion and diuresis.
  Arms: self-posturotherapy

SUMMARY:
The main objective of this study is to evaluate the effectiveness of an auto posturotherapy technique on the RFS at three months of patients treated for lower calyceal urinary stones by extracorporeal lithotripsy (ECL) or retrograde flexible ureteroscopy.

ELIGIBILITY:
pré Inclusion Criteria:

* Patient having read and signed the consent form for participation in the study • Patient candidate for an intervention on a lower calyx stone <15mm by LEC or URSS

Patients meeting all of the following criteria may be definitively included in the study:

* Patient treated by LEC, or patient treated by URSS and for whom the presence of lower calyceal fragments has been observed by endoscopy
* Absence of JJ stent (patients for whom a JJ stent was implanted after URSS or before LEC may be included as soon as it is removed)

Exclusion Criteria:

* Patients presenting one of the following criteria will not be included in the study:

  * Renal or ureteral malformation: ureteral stenosis, pyelo-ureteral junction syndrome, horseshoe kidney, para calyceal diverticulum, pelvic kidney.
  * LEC session interrupted due to treatment intolerance
  * Physical disability making posturotherapy impossible (particularly spinal, etc.), morbid obesity, major gastroesophageal reflux, heart or respiratory failure.
  * Balance disorder which would not allow self-posturotherapy to be carried out alone.
  * Patient under legal protection, under guardianship or under curatorship
  * Posturotherapy carried out while wearing a JJ probe
  * Posturotherapy carried out by a third party (physiotherapist or other)
  * Pregnant or breastfeeding patient
  * Patient not affiliated to the French social security system
  * Impossibility of providing the subject with informed information and/or giving written informed consent: dementia, psychosis, disorders of consciousness, non-French speaking patient
  * Treatment that may modify the clearance of fragments (beta blocker, diuretic, etc.)
  * Patient included in another therapeutic study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
stone free rate | 3 month

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Edouard Herriot -, Lyon
  - Clinique La Croix du Sud, Quint-Fonsegrives

IPD SHARING:
Plan to Share IPD: No